CLINICAL TRIAL: NCT01031602
Title: Assessment of the Prevalence of Sexual Dysfunction, Depression, and Anxiety in Underserved and Minority Patients With Gynecologic Cancers
Brief Title: Assessment of Sexual Dysfunction, Depression and Anxiety in Underserved, Minority Gynecologic Cancers Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0436
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Gynecologic Cancer
Keywords: Cancer; Gynecology; Sexual Dysfunction; Depression; Anxiety; Underserved; Minority; Psychological distress
MeSH Terms: conditions — Neoplasms; Sexual Dysfunction, Physiological; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psych Needs Assessment: Female Sexual Function Index (FSFI), Hospital Anxiety and Depression Scale (HADS), and a demographic questionnaire given to underserved and minority women with a gynecologic cancer or premalignant condition.
  Interventions: Behavioral: Surveys

INTERVENTIONS:
Behavioral: Surveys — Surveys -- Female Sexual Function Index (FSFI), the Hospital Anxiety and Depression Scale (HADS), and a demographic questionnaire completed at time of clinic appointment, taking about 20 minutes.
  Other Names: Questionnaire

SUMMARY:
Objectives:

* Assess the prevalence and severity of depression and anxiety in underserved and minority women seen in the gynecologic oncology clinic at Lyndon Baines Johnson General Hospital.
* Assess the prevalence and severity of sexual dysfunction in this patient population.

DETAILED DESCRIPTION:
The instruments used in this study will be completed at one timepoint, by those women who choose to participate, anonymously. The questionnaires will be preceded with a statement informing the patient that by completing the study questionnaires she is consenting to study participation. No patient names or medical record numbers will be documented.

When a patient checks in for her clinic appointment, she will receive a packet of study materials consisting of a cover letter describing the study objectives, the Female Sexual Function Index, the Hospital Anxiety and Depression Scale, and a demographic questionnaire. The tools used in this study will be available in both English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

- Women seen at the Gynecologic Oncology Clinic at the Lyndon Baines Johnson General Hospital. The women must be able to read and write either English or Spanish.

Exclusion Criteria:

- Women who are unable to complete the questionnaires.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women seen at the Gynecologic Oncology Clinic at the Lyndon Baines Johnson (LBJ) General Hospital and able to read and write either English or Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sexual Dysfunction, Depression, and Anxiety in Patients Surveyed | Survey perfomed at single point in time

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Study Chair — UT MD Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson (LBJ) General Hosptial, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org